CLINICAL TRIAL: NCT05757934
Title: Exploring the Long-term Cardiovascular Effects of Vaping: a Longitudinal Study
Brief Title: Exploring the Long-term Cardiovascular Effects of Vaping
Acronym: LIGER
Status: Active, not recruiting | Type: Observational
Sponsor: Sheffield Hallam University (Other)
Collaborators: Leeds Beckett University (Other)
Responsible Party: Principal Investigator, Markos Klonizakis, Professor of Vascular and Clinical Physiology, Sheffield Hallam University
Other Study IDs: ER49341917
Record Dates: First submitted 2023-02-07; First posted 2023-03-07 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases
Keywords: vaping; macrocirculation; smoking; blood biomarkers
MeSH Terms: conditions — Cardiovascular Diseases; Vaping; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: vapers, who are ex-smokers.
- Group B: vapers with no previous smoking experience.
- Group C: vapers, who are dual users (i.e., those who vape and smoke).
- Group D: ex-smokers who don't vape.

SUMMARY:
Smoking is the "leading, preventable death-cause worldwide", being responsible for almost 700,000 deaths in the E.U. annually. Therefore, implementing successful, long-term smoking cessation strategies is a long-term priority for the NHS.

Recent evidence suggests that e-cigarettes (i.e., vaping) are a successful cessation tool, with around 3.6 million users in the UK. There are concerns about long-term vaping, particularly in relation to their cardiovascular effects, as there are no relevant, longitudinal studies.

Therefore, we propose a 38-month, four-group longitudinal study exploring the cardiovascular physiological effects of the use of e-cigarettes over a two-year period, informing policy makers and e-cigarette users (vapers). Our study was developed with the support of vapers.

The main research question is whether there are any differences in cardiovascular physiology between vapers, who are ex-smokers (Group A), vapers with no previous smoking experience (Group B), dual users (i.e., those who vape and smoke (Group C) and ex-smokers who don't vape (Group D).

Two-hundred participants from Sheffield and Leeds will be invited on five occasions (baseline, as well as 6-,12-,18- and 24-months post-baseline).

We will assess macrovascular and lung function, cardiovascular disease risk (through questionnaires and blood biomarkers), vaping and smoking dependence, smoking and and vaping history among others.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Age ≥18 years of either gender. Specific group inclusion criteria include:

Group A: Ex-smokers with previous smoking history of at least two years, who vape for at least one year, at least 50 puffs a day.

Group B: Current vapers who have been vaping daily (minimum 50 puffs/day) for at least one year, with no previous smoking history, Group C: Current vapers (50 puffs/day), who smoke at least 20 cigarettes per week. Group D: Ex-smokers, who have stopped smoking for a period greater than one year and who currently do not vape.

Exclusion Criteria:

* Non-ambulant people and people with a recent (e.g., within 6 months) CVD event (e.g. stroke, myocardial infarction) or cardiac surgery,
* pregnancy,
* people who require major surgery (which will prevent them of taking part in the study),
* people who are unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vapers conforming to specific group criteria in wider Sheffield and Leeds areas, in the U.K.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Brachial artery FMD using ultrasound | 24 months
  Baseline scanning to assess resting vessel diameter will be recorded over 3 min, following a 10-min resting period. The brachial artery will be imaged at a location 3 to 7 cm above the antecubital crease to create a flow stimulus in the brachial artery. The images will be obtained with a Viamo C100 (Canon Medical Systems Europe B.V., Zoetermeer, Netherlands) unit using a 7.5MHz PSI-30BX (Canon Medical Systems Europe B.V., Zoetermeer, Netherlands) transducer. A sphygmomanometric cuff will be placed on the forearm; the cuff will be inflated at least 50 mmHg above systolic pressure to occlude artery inflow for 5 min. Recordings will commence 30s before cuff deflation and continuing for 3 min after. FMD will be expressed as a change in post-stimulus diameter evaluated as a percentage of the baseline diameter.

SECONDARY OUTCOMES:
Brachial artery FMD using ultrasound | 3 months
  As in 24 months.
Brachial artery FMD using ultrasound | 6 months
  As in 24 months.
Brachial artery FMD using ultrasound | 12 months
  As in 24 months.
Brachial artery FMD using ultrasound | 18 months
  As in 24 months.
Vascular assessment of biomarkers | 24 months
  Venous blood samples (10 ml) will be obtained from the participants via a superficial arm vein to assess C-reactive protein, IL-12 (p70), sICAM-1, IL-8 and vWF.
Vascular assessment of biomarkers | 12 months
  Venous blood samples (10 ml) will be obtained from the participants via a superficial arm vein to assess C-reactive protein, IL-12 (p70), sICAM-1, IL-8 and vWF.
Vascular assessment of biomarkers | 6 months.
  Venous blood samples (10 ml) will be obtained from the participants via a superficial arm vein to assess C-reactive protein, IL-12 (p70), sICAM-1, IL-8 and vWF.
Vascular assessment of biomarkers | 18 months
  Venous blood samples (10 ml) will be obtained from the participants via a superficial arm vein to assess C-reactive protein, IL-12 (p70), sICAM-1, IL-8 and vWF.
Lung function | 24 months
  Lung function including FEV1, FVC and vital capacity will be measured according to international guidelines (ATS/ERS guidelines).
Lung function | 6 months
  Lung function including FEV1, FVC and vital capacity will be measured according to international guidelines (ATS/ERS guidelines).
Lung function | 12 months
  Lung function including FEV1, FVC and vital capacity will be measured according to international guidelines (ATS/ERS guidelines).
Lung function | 18 months
  Lung function including FEV1, FVC and vital capacity will be measured according to international guidelines (ATS/ERS guidelines).
Smoking dependence | baseline
  Using Fagerström questionnaire.
Vaping dependence | baseline
  Using Vaping dependence questionnaire.
Vaping dependence | 6 months
  Using Vaping dependence questionnaire.
Vaping dependence | 12 months
  Using Vaping dependence questionnaire.
Vaping dependence | 18 months
  Using Vaping dependence questionnaire.
Vaping dependence | 24 months
  Using Vaping dependence questionnaire.
Smoking dependence | 24 months
  Using Fagerström questionnaire.
Smoking dependence | 18 months
  Using Fagerström questionnaire.
Smoking dependence | 12 months
  Using Fagerström questionnaire.
Smoking dependence | 6 months
  Using Fagerström questionnaire.
Change in CV risk profile | 24 months
  Q-risk assessment
Change in CV risk profile | 18 months
  Q-risk assessment
Change in CV risk profile | 12 months
  Q-risk assessment
Change in CV risk profile | 6 months
  Q-risk assessment
Anthropometrics | baseline
  height (m), weight (m) to calculate body mass index (BMI) as weight divided by height squared,
Anthropometrics | 24 months
  height (cm), weight (m) to calculate body mass index (BMI) as weight divided by height squared,
Anthropometrics | 18 months
  height (cm), weight (m) to calculate body mass index (BMI) as weight divided by height squared,
Anthropometrics | 12 months
  height (cm), weight (m) to calculate body mass index (BMI) as weight divided by height squared,
Anthropometrics | 6 months
  height (cm), weight (m) to calculate body mass index (BMI) as weight divided by height squared,
Anthropometrics | baseline
  heart rate variability (assessed as normal-to-normal (NN) intervals).
Anthropometrics | baseline
  blood pressure (mmHg).
Anthropometrics | 6 months
  blood pressure (mmHg).
Anthropometrics | 12 months
  blood pressure (mmHg).
Anthropometrics | 18 months
  blood pressure (mmHg).
Anthropometrics | 24 months
  blood pressure (mmHg).
Anthropometrics | 24 months
  heart rate variability (assessed as normal-to-normal (NN) intervals).
Anthropometrics | 18 months
  heart rate variability (assessed as normal-to-normal (NN) intervals).
Anthropometrics | 12 months
  heart rate variability (assessed as normal-to-normal (NN) intervals).
Anthropometrics | 6 months
  heart rate variability (assessed as normal-to-normal (NN) intervals).
Smoking abstinence | 24 months
  For Groups A, B and D smoking abstinence will be defined by the presence of CO < 10ppm
Smoking abstinence | 18 months
  For Groups A, B and D smoking abstinence will be defined by the presence of CO < 10ppm
Smoking abstinence | 12 months
  For Groups A, B and D smoking abstinence will be defined by the presence of CO < 10ppm
Smoking abstinence | 6 months
  For Groups A, B and D smoking abstinence will be defined by the presence of CO < 10ppm

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Hallam University, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided